CLINICAL TRIAL: NCT00884871
Title: A Prospective Cohort Study of the Impact of Surgically-Induced Weight Loss on Pelvic Floor Disorders
Brief Title: Study of Surgically-Induced Weight Loss on Pelvic Floor Disorders
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Emily L. Whitcomb, University of California San Diego
Other Study IDs: 071113
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor disorders; weight loss
MeSH Terms: conditions — Pelvic Floor Disorders; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic adjustable gastric banding: 100 obese women undergoing laparoscopic adjustable gastric banding
  Interventions: Procedure: LapBand

INTERVENTIONS:
Procedure: LapBand — Prospective observation study of 100 obese women undergoing laparoscopic gastric banding to determine impact of weight loss on pelvic floor disorders

SUMMARY:
The specific aim of this study is to evaluate the effect of surgically-induced weight reduction, as achieved by laparoscopic gastric banding or sleeve gastrectomy, on pelvic floor disorders such as stress urinary incontinence, overactive bladder, anal incontinence, and pelvic organ prolapse in severely, morbidly and super-obese women using a prospective, observational study design.

ELIGIBILITY:
Inclusion Criteria:

* surgical eligibility met by Center for the Treatment Obesity criteria
* morbid obesity (BMI > 40 kg/m2) or severe obesity (BMI > 33 kg/m2) in presence of NIH co-morbidities
* willing to participate in study, including completion of self-reported questionnaires

Exclusion Criteria:

* pregnancy or planned pregnancy
* recent pregnancy or pelvic surgery
* age < 21 years
* known neurologic disease or pelvic pathology

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 obese women who have met surgical eligibility for laparoscopic adjustable gastric banding at the Center for the Treatment of Obesity at UCSD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of pelvic floor disorders ascertained by Epidemiology of Prolapse and Incontinence Questionnaire | 12 months

SECONDARY OUTCOMES:
Weekly incontinence episodes and pad use ascertained by incontinence diary | 12 months
Quality of life impact ascertained by validated measures (PFIQ, PFDI, FISI, and PGI-I) | 12 months
Sexual function ascertained by validated measure (PISQ) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Whitcomb, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Medical Center, La Jolla, California, United States